CLINICAL TRIAL: NCT05942040
Title: Translating Data Science to Palliative Care Practice for Persons Living With Dementia
Brief Title: Translating Data Science to Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elizabeth A. Luth, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro2023000794; P30AG064105 (NIH)
Record Dates: First submitted 2023-06-22; First posted 2023-07-12 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease and Related Dementias
Keywords: Palliative care; Community based palliative care; Family care partner; Algorithm
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group will consist of all MA plan members eligible for community-based palliative care and of those who refused it (to calculate refusal rate) during the six month period following the introduction of tailored informational materials developed on CBPC
  Interventions: Other: Tailored Palliative Care Information
- Control Group (No Intervention): Control group will be a retrospective review of individuals who were eligible for community-based palliative care and of those who refused it, for the 6-month period prior to introducing the tailored informational materials. All of these individuals will have received usual care/information regarding community-based palliative care.

INTERVENTIONS:
Other: Tailored Palliative Care Information — This study test feasibility and acceptability of implementing tailored informational materials into clinician's discussions about CBPC with MA plan members who are eligible for the service.
  Arms: Intervention Group

SUMMARY:
This research study is intended to 1) better understand seriously ill adults' and their family care partners' (FCP), particularly for persons living with dementia (PLwD), barriers to accepting community-based palliative care (CBPC); 2) develop an intervention to address barriers; and 3) pilot test whether the intervention has an impact on CBPC uptake. The intervention will consist of 1) a set of informational material describing the benefits of CBPC for the CBPC team to use when presenting CBPC to members of a Medicare Advantage plan and their FCP; and 2) processes for tailoring information delivery so that eligible members and their FCP receive information about CBPC that reflects their individualized risk as identified by the Medicare Advantage program's validated 12-month mortality risk algorithm.

The clinical trial portion of the study refers to the pilot test (Aim 3 as described below).

DETAILED DESCRIPTION:
Aim 1. Engage Family Care Partners (FCPs) and Community Based Palliative Care (CBPC) team members to identify barriers to CBPC. Aim 1 will incorporate the perspectives of CBPC team members and Medicare Advantage (MA) plan members and FCPs of person living with dementia (PLwD) and those with other diagnoses who refused CBPC services. Aim 2. Develop and obtain feedback on a) informational materials for CBPC team members to use when speaking with MA members and FCPs about CBPC and b) processes for tailoring information delivery based on a members's algorithm-identified risk profile. Most participants will be recruited from Aim 1 participants. Additional participants will be recruited as necessary. Aim 3. Conduct a pre-post trial to determine the feasibility and acceptability of the materials and using them in existing clinical workflows for their a) impact on CBPC enrollment for CBPC-eligible individuals, including PLwD, and b) end-user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* VNS Health Total Medicare Advantage Plan member
* identified as eligible for community-based palliative care by the VNS Health Total palliative care team during the study period (6-month period prior to introduction of the intervention and the 6-month period following the intervention)
* 18 years of age or older

Exclusion Criteria:

* non-VNS Health Total Medicare Advantage Plan member
* VNS Health Total plan members not identified as eligible for community-based palliative care by the palliative care team during the study period (6-month period prior to introduction of the intervention and the 6-month period following the intervention)
* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Luth, PhD, Principal Investigator — Rutgers University
Locations (1):
- VNS Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 301 individuals enrolled in the study. 294 participants enrolled via a waiver of consent to retrospectively analyze electronic records (primary outcome only). Of these, 111 were in intervention; 182 in control. 7 participants were palliative care team members who provided satisfaction data (secondary outcome only). Of these 7, 1 individual dropped out of the study after consent and prior to providing any data. Reported results are based on 300 participants for whom data were provided.
Groups:
- Intervention Group: Intervention group will consist of all MA plan members eligible for community-based palliative care and of those who refused it (to calculate refusal rate) during the six month period following the introduction of tailored informational materials developed on CBPC.
  Note: Post-intervention planned to be 6 months, in implementation was 5-months due to delayed initiation of intervention.
- Control Group: Control group will be a retrospective review of individuals who were eligible for community-based palliative care and of those who refused it, for the 6-month period prior to introducing the tailored informational materials. All of these individuals will have received usual care/information regarding community-based palliative care.
  Note: Pre-intervention planned to be 6 months, in implementation was 5-months due to delayed initiation of intervention.
- Community Based Palliative Care Team Members: Tailored Palliative Care Information: This study test feasibility and acceptability of implementing tailored informational materials into clinician's discussions about CBPC with MA plan members who are eligible for the service.
  Note: Post-intervention planned to be 6 months, in implementation was 5-months due to delayed initiation of intervention.
Period: Overall Study
Arm/Group | Intervention Group | Control Group | Community Based Palliative Care Team Members
Started | 111 | 182 | 7
Completed | 111 | 182 | 4
Not Completed | 0 | 0 | 3
Not completed — No longer employed at study site. | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Community Based Palliative Care Team Members | Total
Number analyzed (Participants) | 111 | 182 | 7 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.7 (10.7) | 86.5 (11.1) | 50.1 (12.6) | 84.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 130 | 7 | 226
  Male | 22 | 52 | 0 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 79 | 1 | 118
  Not Hispanic or Latino | 0 | 0 | 6 | 6
  Unknown or Not Reported | 73 | 103 | 0 | 176
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 0 | 5
  Asian | 14 | 13 | 0 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 33 | 58 | 4 | 95
  White | 36 | 80 | 2 | 118
  More than one race | 6 | 8 | 0 | 14
  Unknown or Not Reported | 21 | 19 | 1 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 111 | 182 | 7 | 300
Palliative care refusal rate [Count of Participants; unit: Participants] — Population: This measure was assessed for intervention and control group participants only. community palliative care team members did not complete it.
  Participants
    number analyzed (Participants) | 111 | 182 | 0 | 293
    Enrolled in Palliative Care | 50 | 69 |  | 119
    Declined Palliative Care | 61 | 113 |  | 174
    Did not contribute data | 0 | 0 |  | 0
End-User Satisfaction Survey [Mean (Standard Deviation); unit: units on a scale] — End-User Satisfaction was assessed using The Measurement of End-User Computing Satisfaction 12-item survey (Doll & Torkzadeh (1988). This survey assesses satisfaction with an information system related to accuracy, format, ease of use, and timeliness. Each item is rated 1-5, with higher scores representing more positive ratings. Total minimum score=12 (lowest satisfaction), maximum score=60 (highest satisfaction). Population: This feasibility and acceptability measure was only assessed for community based palliative care team members. It was not assessed for intervention and control group participants.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 7 | 7
    (all) |  |  | 35.4 (5.7) | 35.4 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Palliative Care Refusal Rate
Description: The investigators will assess refusal rate using the MA plan's electronic health records. Refusal rate will be calculated as # of eligible individuals refusing palliative care / total # of individuals eligible for palliative care
Time Frame: Baseline through 10 months. Pre (control group) test for 5 months prior to intervention. Post (intervention group) for 5 months during intervention.
Population: All participants who were eligible for the VNS Health Total Medicare Advantage plan's community-based palliative care program in the 5 months pre-intervention or 5-months post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 111 | 182
Participants
  Enrolled in Palliative Care | 50 | 69
  Declined Palliative Care | 61 | 113
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other — Pre-post test; p = 0.17, Regression, Logistic; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.43 to 1.16], Standard Error of Mean 0.18

2. Secondary Outcome: CBPC Team Members Satisfaction
Description: Investigators will assess intervention feasibility and acceptability using the end-user satisfaction survey. End-User Satisfaction ratings for each concept are scored as 1 (almost never); 2 (some of the time); 3 (about half the time); 4 (most of the time); 5 (almost always). Minimum score is 12; maximum 60, with higher scores indicating greater satisfaction.
Time Frame: Baseline, 2.5 and 5 months into intervention delivery.
Population: All CBPC Team Member participants who provided survey responses to the End-User Satisfaction survey at 2.5 and 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Based Palliative Care Team Members
Number analyzed (Participants) | 4
score on a scale
  Baseline | 35 (5.7)
  2.5 months | 47.5 (9.7)
  5 months | 52 (11.8)

ADVERSE EVENTS:
Time Frame: Primary outcome: Electronic record data were retrospectively analyzed via waiver of consent for 294 individuals from 12/1/23-9/30/24. Although we initially planned for two 6-month periods, in implementation we conducted the intervention over two 5-month periods (5 months pre-intervention and 5 months post-intervention). Secondary outcome: We collected feasibility data from 7 palliative care team members from 2/14/24-9/30/24 who consented. Study start now reflects date of team member consent.
Groups:
- Community Based Pallaitve Care Team Members: Tailored Palliative Care Information: This study test feasibility and acceptability of implementing tailored informational materials into clinician's discussions about CBPC with MA plan members who are eligible for the service.
  Note: Post-intervention planned to be 6 months, in implementation was 5-months due to delayed initiation of intervention.
Arm/Group | Intervention Group | Control Group | Community Based Pallaitve Care Team Members
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/182 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/182 | 0/7
Other Adverse Events (participants affected / at risk) | 0/111 | 0/182 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT05942040/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT05942040/ICF_001.pdf